CLINICAL TRIAL: NCT00850746
Title: A Phase 1, Randomized, Double-Blind, Placebo- and Active- Controlled, Crossover Study to Evaluate the Effect of Repeat Oral Doses of YM443 on Cardiac Repolarization in Healthy Male and Female Adult Subjects
Brief Title: A Study to Evaluate the Effect of Repeat Oral Doses of YM443 on Cardiac Repolarization in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Astellas Pharma Inc (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple
Other Study IDs: 443-CL-048
Record Dates: First submitted 2009-02-23; First posted 2009-02-25 (Estimated); Last update posted 2014-03-24 (Estimated); Status verified 2014-03

CONDITIONS: Functional Dyspepsia
Keywords: QT interval; Cardiac Repolarization; Cardiac Conduction; Healthy Subjects; YM443 (Z-338, acotiamide hydrochloride); Evaluation of QT Interval
MeSH Terms: interventions — Z 338; Moxifloxacin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- A. Placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- B. Ym443 Lower Dose (Experimental)
  Interventions: Drug: YM443
- C. YM443 Higher Dose (Experimental)
  Interventions: Drug: YM443
- D. Moxiflocxacin (Active Comparator)
  Interventions: Drug: Moxifloxacin

INTERVENTIONS:
Drug: YM443 — Oral
  Other Names: Z-338; acotiamide hydrochloride
  Arms: B. Ym443 Lower Dose; C. YM443 Higher Dose
Drug: Placebo — Oral
  Arms: A. Placebo
Drug: Moxifloxacin — Oral
  Other Names: Avelox
  Arms: D. Moxiflocxacin

SUMMARY:
This study evaluates whether YM443 causes any changes in the electrocardiogram of healthy adults.

DETAILED DESCRIPTION:
Each subject participates in all four treatment periods separated by washout periods.

In order to maintain the blind between arms, all subjects will receive the same number of tablets per day in each period of either active drug or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Healthy Male or non pregnant, non lactating female
* Weighing at least 45 kg
* Body Mass Index (BMI) between 18 and 32 kg/m2

Exclusion Criteria:

* The subject has evidence of any cardiac conduction abnormalities
* The subject has a previous history of any medical or psychiatric condition that would preclude participation in the study
* The subject has participated in another clinical trial in the last 30 days
* The subject anticipates an inability to abstain from alcohol, or caffeine use, or from grapefruit and grapefruit juice from 48 hours prior to the administration of the first dose of YM443 on Day 1 of Period 1 and throughout the duration of the study
* The subject has used tobacco-containing products and nicotine or nicotine-containing products within six months prior to Screening
* The subject consumes more than 5 units of alcoholic beverages (one unit is 12 ounces of beer, 4 ounces of wine or 1 ounce of spirits) per week or has a history of substance abuse, drug addiction, or alcoholism within 2 years prior to Screening
* The subject has donated any whole blood or cellular blood component or has undergone significant loss of blood or has received transfusion of any blood or blood products within 56 days of Day -1 of Period 1 or has donated plasma within 7 days of Day -1 of Period 1

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 80 (Actual)
Dates: Start 2009-02; Primary Completion 2009-04 (Actual); Study Completion 2009-04 (Actual)

PRIMARY OUTCOMES:
Mean change in the QTcF (Fridericia's correction) between each active treatment and placebo | Following four days of dosing

SECONDARY OUTCOMES:
The mean change of the QTcI (Individual correction) and QTcB (Bazett's correction) between each active treatment and placebo. | Following four days of dosing
The pharmacokinetics of YM443 in these subjects | Day 5
The safety and tolerability of YM443 | Following four days of dosing

CONTACTS AND LOCATIONS:
Overall Officials: Use Central Contact, Study Director — Astellas Pharma Global Development
Locations (1):
- Tacoma, Washington, United States